CLINICAL TRIAL: NCT06743165
Title: New Generation Rehabilitation Approach in Children With Dysfunctional Voiding: Pelvic Floor Muscle Training and Dynamic Neuromuscular Stabilization Training With Transabdominal Ultrasound, a Randomized Controlled Trial
Brief Title: New Generation Rehabilitation Approach in Children With Dysfunctional Voiding
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir University of Economics (Other)
Collaborators: Health Institutes of Turkey (Other Government)
Responsible Party: Principal Investigator, Seda Yakit Yesilyurt, Assist. Prof., Izmir University of Economics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYY_IEU_4
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Dysfunctional Voiding; Children; Pelvic Floor Muscle Training; Ultrasound; DNS

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DNS Group (Experimental): This group includes 18 children with Dysfunctional voiding, aged between 6 and 14 years.
  Interventions: Behavioral: Pelvic floor muscle training with ultrasound biofeedback; Behavioral: Dynamic neuromuscular stabilization exercise
- Standard exercise group (Active Comparator): This group includes 18 children with Dysfunctional voiding, aged between 6 and 14 years.
  Interventions: Behavioral: Pelvic floor muscle training with ultrasound biofeedback

INTERVENTIONS:
Behavioral: Pelvic floor muscle training with ultrasound biofeedback — Pelvic floor muscle training (PFMT) will be given to both groups with transabdominal US. PFMT will be applied by physiotherapists who have received training and supervision from physiotherapists who are experts in the field of pelvic floor US imaging and pelvic floor muscle training with US. Pelvic floor muscle training will be applied with a GE Brand LOGIQ P8 model transabdominal ultrasound (GE HealthCare) US device under the supervision of an expert physiotherapist. Parents and children will be informed about PFMT.
Behavioral: Dynamic neuromuscular stabilization exercise — Dynamic neuromuscular exercises (DNS) involve the joint activation of the intrinsic muscle group of the spine, which includes the cervical flexors and extensors, diaphragm, transversus abdominis, multifidus and pelvic floor, which form the integrated spinal stabilization system. The application principles are joint centering, core stabilization - Integrated spinal stabilization system and stabilization function of the diaphragm. DNS training will be applied in three stages. Preparation for exercises, IAB regulation and application of exercises according to developmental kinesiology positions. Exercises will start with preparatory training. In preparatory training, stroking, brushing and tapping techniques will be taught and self-facilitation will be demonstrated in order to increase proprioceptive input to the lower extremity, upper extremity, trunk and pelvic region. Fascial mobilizations will be performed to the foot and hand regions.
  Arms: DNS Group

SUMMARY:
The investigators hypothesize that Dynamic Neuromuscular Stabilization training, a next-generation exercise approach, and transabdominal ultrasound-guided pelvic floor muscle training (PFMT) will be more effective than PFMT guided solely by transabdominal ultrasound in reducing post-void residual volume, improving voiding disorder symptoms, and enhancing pelvic floor muscle relaxation in children with dysfunctional voiding.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-14 years,
* Diagnosed with dysfunctional urination according to uroflowmetry measurement results and clinical examination findings,
* Children who consent to participate in the study with the consent of their mother, father or legal guardian (legal representative) will be included in the study.

Exclusion criteria:

* Children under 6 years of age,
* Those with anatomical changes in the urinary system,
* Those with spina bifida,
* Those with a history of active urinary tract infection,
* Those with a neurological disease,
* Those with accompanying respiratory system disease,
* Those with cognitive impairment,
* Those with mental retardation,
* Children whose bladder image is unclear in the pelvic floor evaluation with US,
* Children who have previously undergone orthopedic surgery will not be included in the study.

PS:

* Children who cannot comply with the application of pelvic floor muscle training,
* Children who have missed 2 or more sessions of the treatment program will be excluded from the study.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-02-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the amount of post-void residue | From enrollment to the end of treatment at 8 weeks
  After EMG-Uroflowmetry test: Post-void residual measurement will be made by transabdominal ultrasound 5 minutes after voiding. In repeated measurements, the amount of urine remaining in the bladder of 20 ml or more will be considered pathological.
Change in EMG-Uroflowmetry measurements-peak flow rate | From enrollment to the end of treatment at 8 weeks
  EMG-Uroflowmetry test procedure: Before the test, the device will be calibrated and the scale of the interpretation sheet will be set to 1:1 for flow rate (ml/sec) and time (sec). The test will be performed in a quiet and private room and the patient will be asked to drink as much fluid as the expected bladder capacity ((age in years+1)x30) 1 hour before the test. During the test, the EMG activity of the pelvic floor muscles will also be evaluated. Voided volume (ml), peak flow rate (Q max, ml/sec) and uroflow curve interpretation will also be used. Those with decreased flow rate and stacco/interminant flow pattern will be considered pathological.
Change in EMG-Uroflowmetry measurements-Pelvic Floor EMG activity | From enrollment to the end of treatment at 8 weeks
  EMG-Uroflowmetry test procedure: Before the test, the device will be calibrated and the scale of the interpretation sheet will be set to 1:1 for flow rate (ml/sec) and time (sec). The test will be performed in a quiet and private room and the patient will be asked to drink as much fluid as the expected bladder capacity ((age in years+1)x30) 1 hour before the test. During the test, the EMG activity of the pelvic floor muscles will also be evaluated. Recorded as (µV).

SECONDARY OUTCOMES:
Change in EMG-Uroflowmetry measurements-uroflow curve | From enrollment to the end of treatment at 8 week
  EMG-Uroflowmetry test procedure: Before the test, the device will be calibrated and the scale of the interpretation sheet will be set to 1:1 for flow rate (ml/sec) and time (sec). The test will be performed in a quiet and private room and the patient will be asked to drink as much fluid as the expected bladder capacity ((age in years+1)x30) 1 hour before the test. During the test, the EMG activity of the pelvic floor muscles will also be evaluated. Voided volume (ml), peak flow rate (Q max, ml/sec) and uroflow curve interpretation will also be used. Those with decreased flow rate and stacco/interminant flow pattern will be considered pathological.
Change in EMG-Uroflowmetry measurements - Voided volume | From enrollment to the end of treatment at 8 weeks
  EMG-Uroflowmetry test procedure: Before the test, the device will be calibrated and the scale of the interpretation sheet will be set to 1:1 for flow rate (ml/sec) and time (sec). The test will be performed in a quiet and private room and the patient will be asked to drink as much fluid as the expected bladder capacity ((age in years+1)x30) 1 hour before the test. During the test, the EMG activity of the pelvic floor muscles will also be evaluated. Voided volume (ml), peak flow rate (Q max, ml/sec) and uroflow curve interpretation will also be used. Those with decreased flow rate and stacco/interminant flow pattern will be considered pathological.
Pelvic floor muscle assessment with ultrasound - maximum displacement (cm) | From enrollment to the end of treatment at 8 weeks
  Assessment procedure: Pelvic floor assessment will be performed with transabdominal US. In order for imaging to be performed properly during ultrasound measurement, the child will be asked to consume 250 ml of a caffeine-free liquid before measurement. The measurement will be performed in the lying position with a 2-5 MHz GE Brand LOGIQ P8 model transabdominal ultrasound (GE HealthCare) device in accordance with the protocols in Bo and Bower's studies. In this measurement, a fixed point will be determined at the base of the bladder and the displacement of this fixed point will be taken as basis during pelvic floor muscle assessment.
Pelvic floor muscle assessment with ultrasound - coordination amplitude (cm) | From enrollment to the end of treatment at 8 weeks
  Assessment procedure: Pelvic floor assessment will be performed with transabdominal US. In order for imaging to be performed properly during ultrasound measurement, the child will be asked to consume 250 ml of a caffeine-free liquid before measurement. The measurement will be performed in the lying position with a 2-5 MHz GE Brand LOGIQ P8 model transabdominal ultrasound (GE HealthCare) device in accordance with the protocols in Bo and Bower's studies. In this measurement, a fixed point will be determined at the base of the bladder and the displacement of this fixed point will be taken as basis during pelvic floor muscle assessment.
Pelvic floor muscle assessment with ultrasound - endurance amplitude (%) | From enrollment to the end of treatment at 8 weeks
  Assessment procedure: Pelvic floor assessment will be performed with transabdominal US. In order for imaging to be performed properly during ultrasound measurement, the child will be asked to consume 250 ml of a caffeine-free liquid before measurement. The measurement will be performed in the lying position with a 2-5 MHz GE Brand LOGIQ P8 model transabdominal ultrasound (GE HealthCare) device in accordance with the protocols in Bo and Bower's studies. In this measurement, a fixed point will be determined at the base of the bladder and the displacement of this fixed point will be taken as basis during pelvic floor muscle assessment.
Gross Motor Development Stages | at baseline
  Children's gross motor development stages will be questioned in accordance with the protocol determined by the World Health Organization. The children's time to sit without support, stand with support, crawl, walk with help, stand alone and walk alone will be noted in months.
Change in symptom severity | From enrollment to the end of treatment at 8 weeks
  The severity of children's voiding disorder symptoms will be assessed with the Voiding Disorders Symptom Score. The Voiding Disorders Symptom Score was developed by Akbal et al in 2005 and consists of a total of 14 questions. The 13 questions of the questionnaire evaluate symptoms related to daytime urinary incontinence, symptoms related to nighttime urinary incontinence, frequency of urination in a day, presence of constipation and various symptoms related to urinary incontinence.
Change in symptom severity | 6 months after treatment
  The severity of children's voiding disorder symptoms will be assessed with the Voiding Disorders Symptom Score. The Voiding Disorders Symptom Score was developed by Akbal et al in 2005 and consists of a total of 14 questions. The 13 questions of the questionnaire evaluate symptoms related to daytime urinary incontinence, symptoms related to nighttime urinary incontinence, frequency of urination in a day, presence of constipation and various symptoms related to urinary incontinence.
Pelvic floor muscle assessment with ultrasound - maximum displacement (cm) | 6 months after treatment
  Assessment procedure: Pelvic floor assessment will be performed with transabdominal US. In order for imaging to be performed properly during ultrasound measurement, the child will be asked to consume 250 ml of a caffeine-free liquid before measurement. The measurement will be performed in the lying position with a 2-5 MHz GE Brand LOGIQ P8 model transabdominal ultrasound (GE HealthCare) device in accordance with the protocols in Bo and Bower's studies. In this measurement, a fixed point will be determined at the base of the bladder and the displacement of this fixed point will be taken as basis during pelvic floor muscle assessment.
Pelvic floor muscle assessment with ultrasound - coordination amplitude (cm) | 6 months after treatment
  Assessment procedure: Pelvic floor assessment will be performed with transabdominal US. In order for imaging to be performed properly during ultrasound measurement, the child will be asked to consume 250 ml of a caffeine-free liquid before measurement. The measurement will be performed in the lying position with a 2-5 MHz GE Brand LOGIQ P8 model transabdominal ultrasound (GE HealthCare) device in accordance with the protocols in Bo and Bower's studies. In this measurement, a fixed point will be determined at the base of the bladder and the displacement of this fixed point will be taken as basis during pelvic floor muscle assessment.
Pelvic floor muscle assessment with ultrasound - endurance amplitude (%) | 6 months after treatment
  Assessment procedure: Pelvic floor assessment will be performed with transabdominal US. In order for imaging to be performed properly during ultrasound measurement, the child will be asked to consume 250 ml of a caffeine-free liquid before measurement. The measurement will be performed in the lying position with a 2-5 MHz GE Brand LOGIQ P8 model transabdominal ultrasound (GE HealthCare) device in accordance with the protocols in Bo and Bower's studies. In this measurement, a fixed point will be determined at the base of the bladder and the displacement of this fixed point will be taken as basis during pelvic floor muscle assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Yakıt Yeşilyurt, Asst. Prof., Principal Investigator — Izmir University of Economics
Locations (1):
- Izmir University of Economics, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since no consent has been received from the institutions supporting this project to share the data with third parties, it will not be shared.